CLINICAL TRIAL: NCT06297746
Title: Comparison of Early Outcomes of Primary Total Knee Arthroplasties Performed Using Subvastus and Medial Parapatellar Approaches and Evaluation of Quadriceps Muscle Elastography
Brief Title: Subvastus vs. Medial Parapatellar Approaches in Total Knee Arthroplasty With Quadriceps Muscle Elastography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Mete Ozer, Research Assistant, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: am7mi3VB
Record Dates: First submitted 2024-03-01; First posted 2024-03-07 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Total Knee Arthroplasty
Keywords: Total Knee Arthroplasty; Subvastus Approach; Medial Parapatellar Approach; Shear Wave Elastography; Elastography; Young's Modulus

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Subvastus approach (Active Comparator): Patients indicated for total knee arthroplasty.
  Interventions: Procedure: Subvastus approach
- Medial Parapatellar approach (Active Comparator): Patients indicated for total knee arthroplasty.
  Interventions: Procedure: Medial Parapatellar approach

INTERVENTIONS:
Procedure: Subvastus approach — Subvastus approach
  Arms: Subvastus approach
Procedure: Medial Parapatellar approach — Medial Parapatellar approach
  Arms: Medial Parapatellar approach

SUMMARY:
ABSTRACT

INTRODUCTION

Knee osteoarthritis is a common joint pathology causing joint pain and ambulatory limitations. In primary total knee arthroplasty (TKA) surgeries, medial parapatellar (MP) and subvastus (SV) approaches are frequently used. The MP approach provides good exposure and is more widely used. In the SV approach, the vastus medialis muscle is preserved. Some argue that the extensor mechanism may heal earlier with the SV approach. In this study, unlike previous studies, the investigators aimed to quantitatively compare the early outcomes of MP and SV approaches, through shear wave elastography (SWE) measurements isolated over the vastus medialis and vastus lateralis muscles.

MATERIALS AND METHODS

The study included 20 patients with indications for TKA due to primary osteoarthritis, divided into MP and SV groups. SWE measurements of the vastus medialis and vastus lateralis muscles were performed preoperatively and at 3-month follow-up. Clinical scores (Knee Society Score and WOMAC) and straight leg raising time were recorded both preoperatively and postoperatively.

ELIGIBILITY:
Eligibility Criteria:

Inclusion Criteria:

- Diagnosis of primary osteoarthritis

Exclusion Criteria:

* Diagnosis of secondary osteoarthritis
* Uncontrolled diabetes
* Uncontrolled hypertension

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-07-10 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Shear wave values | 3 month
  Ultrasonic measurements

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Fatih Güven, Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University - Cerrahpasa, Cerrahpasa Faculty of Medicine, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
All demographic data, clinical scores, and elastography measurement results will be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Background] Shinohara M, Sabra K, Gennisson JL, Fink M, Tanter M. Real-time visualization of muscle stiffness distribution with ultrasound shear wave imaging during muscle contraction. Muscle Nerve. 2010 Sep;42(3):438-41. doi: 10.1002/mus.21723. PMID 20665510
- [Background] Dutka J, Skowronek M, Sosin P, Skowronek P. Subvastus and medial parapatellar approaches in TKA: comparison of functional results. Orthopedics. 2011 Jun 14;34(6):148. doi: 10.3928/01477447-20110427-05. PMID 21667899
- [Background] Vaishya R, Vijay V, Demesugh DM, Agarwal AK. Surgical approaches for total knee arthroplasty. J Clin Orthop Trauma. 2016 Apr-Jun;7(2):71-9. doi: 10.1016/j.jcot.2015.11.003. Epub 2015 Dec 3. PMID 27182142
- [Derived] Guven MF, Ozer M, Ozsahin MK, Deger GU, Adaletli I, Aykan Kargin O, Kaynak G, Botanlioglu H. Comparison of early outcomes of primary total knee arthroplasties performed using subvastus and medial parapatellar approaches and evaluation of quadriceps muscle elastography. Arch Orthop Trauma Surg. 2024 Nov;144(11):4839-4847. doi: 10.1007/s00402-024-05570-5. Epub 2024 Sep 23. PMID 39311941